CLINICAL TRIAL: NCT01085500
Title: Mastery Learning Totally Extraperitoneal Inguinal Hernia Repair: Linking Surgical Simulation to Patient Level Outcomes
Brief Title: Mastery Learning Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, David R. Farley, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 09-008118; 1UL1RR024150 (NIH)
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Inguinal Hernia
Keywords: laparoscopic; totally extraperitoneal inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simulation Curriculum (Experimental): General surgery residents will undergo a simulation-based educational curriculum (Mastery Learning TEP Curriculum) on TEP hernia repair
  Interventions: Behavioral: Mastery Learning TEP Curriculum
- Current Practice (Other): General surgery residents will undergo current practice of learning how to perform the TEP repair in the operating room under direct supervision of the staff surgeon without any simulation pre-training.
  Interventions: Procedure: Current Practice

INTERVENTIONS:
Behavioral: Mastery Learning TEP Curriculum — A simulation-based educational curriculum
  Other Names: TEP Curriculum
  Arms: Simulation Curriculum
Procedure: Current Practice — The current practice of learning how to perform the TEP repair in the operating room is under direct supervision of the staff surgeon without any simulation pre-training.
  Arms: Current Practice

SUMMARY:
Abstract: Minimally invasive techniques are now ubiquitous in the management of surgical disease. Competence in laparoscopy requires specialized training and practice. With the decrease of resident work hours, training programs need to explore and adopt efficient strategies to teach and evaluate laparoscopic skills. For economic, ethical, and legal considerations, the operating room may no longer be the ideal environment for teaching these basic technical skills. There appears to be a role for simulation in response to this need. The transfer of laparoscopic skills learned in a simulated environment to the operating room has showed mixed results. Overall, it seems that surgical skills training outside the operating room is beneficial, but the best method(s) of designing, implementing and evaluating such skills curriculums have yet to be identified.

The laparoscopic totally extraperitoneal (TEP) inguinal hernia repair is an example of a procedure that is associated with a steep learning curve and requires mastery of basic laparoscopic skills. In addition, an increased recurrence and complication rates in the early learning curve of this procedure, underscores the importance of adequate training. The current practice of teaching the TEP repair in the operating room under an apprenticeship-based model is associated with increased operative time and costs. We propose that the training of surgical trainees outside the operating room with a structured, mastery oriented simulation-based curriculum will help reduce the learning curve of the TEP repair, improve operative performance, and decrease operative time and costs.

DETAILED DESCRIPTION:
Specific Aims:

Inguinal hernias are a common ailment of the general population. Their surgical management through a laparoscopic totally extraperitoneal (TEP) approach has been shown to lead to less discomfort and faster recovery than do classic open repairs with equal effectiveness. Nonetheless, the TEP repair has not been adopted widely because of concerns regarding a substantial learning curve. In addition, the current practice of teaching the TEP procedure in the operating room under an apprenticeship-based model is associated with increased operative time and cost. The training of surgeons in laparoscopic skills outside the operating room with simulation-based strategies has emerged as an attractive alternative. Many studies have demonstrated that trainees who practice laparoscopic skills in a simulated environment show improvement of those skills when tested in that same environment. Few studies however, have been able to demonstrate a direct correlation between such simulation training and improved performance in the operating room. It appears from these studies that surgical skills training outside the operating room is beneficial, but the best methods have yet to be identified.

Our long-term research goal is to explore and adopt efficient simulation-based strategies to teach and evaluate surgical skills to surgical trainees. Our objective for this study is to design and evaluate a simulation-based curriculum based upon the concepts of mastery learning theory (achievement of pre-specified expert-derived benchmarks without time constraints) and to develop an objective mean of assessing operative performance that will both aid in shortening the learning curve of the TEP inguinal hernia repair for surgical trainees. Our central hypothesis is that the training of surgery residents outside the operative room with simulation-based strategies, such as the TEP mastery learning curriculum will improve operative performance and reduce operative time during the TEP repair. The rationale for this study is that the identification of effective strategies to shorten the learning curve of the TEP repair that translate into decreased operative time will not only increase the adoption of the TEP repair with its inherent benefits to more candidate patients, but will also lead to substantial cost-savings and perhaps improved patient outcomes. We are especially well prepared to complete this study as we are a part of an academic referral center that treats a myriad of inguinal hernias patients and educates hundreds of surgical residents on a continuous basis.

Specific Aim 1: To compare the TEP mastery learning curriculum with the apprenticeship-based model of learning the TEP repair in the operative room on operative time and operative performance of TEP inguinal hernia repairs performed by surgical trainees.

Hypothesis 1a: Surgical trainees who undergo the TEP mastery learning curriculum will achieve lesser mean operative times while performing a TEP inguinal hernia repair when compared to those who followed the apprenticeship-based model.

Hypothesis 1b: Surgical trainees who undergo the TEP mastery learning curriculum will achieve greater mean operative performance scores while performing a TEP inguinal hernia repair when compared to those who followed the apprenticeship-based model.

Secondary Aim:

Compare the rate of TEP inguinal hernia repair post-operative complications, specifically urinary retention for patients operated on by surgical residents who underwent the mastery learning curriculum versus those who underwent the apprenticeship-based model.

This research is innovative because it will challenge the current paradigm of teaching basic laparoscopic skills in the operative room and will strive to link surgical education methods to objective patient level outcomes such as operative time and cost. At the completion of this project, it is our expectation that we will be better prepared to continue our efforts of translating new educational modalities/technologies to improve the delivery of healthcare. Our anticipated findings will have a relevant impact in how we educate the surgeons of tomorrow.

ELIGIBILITY:
Inclusion Criteria:

* General surgery residents (male or female), regardless of age or previous laparoscopic experience, who are able to perform at least 2 TEP inguinal hernia repairs during the study period (January - December 2010)
* Postgraduate Year (PGY) 1 to PGY 5 general surgery residents.
* Have the procedure supervised by one of the following expert laparoscopic surgeons: Dr. David Farley, Dr. Bingener-Casey, Dr. Swain, Dr. Kendrick

Exclusion Criteria:

- PGY 1 designated preliminary residents (Urology, Orthopedics, Neurosurgery and Anesthesia) or PGY 1 non-designated preliminary residents who are applying to fields other than general surgery.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Farley, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Zendejas B, Cook DA, Bingener J, Huebner M, Dunn WF, Sarr MG, Farley DR. Simulation-based mastery learning improves patient outcomes in laparoscopic inguinal hernia repair: a randomized controlled trial. Ann Surg. 2011 Sep;254(3):502-9; discussion 509-11. doi: 10.1097/SLA.0b013e31822c6994. PMID 21865947

RESULTS

PARTICIPANT FLOW:
Recruitment Details: General surgery residents were recruited from the Mayo Clinic, Rochester, Minnesota from January to September 2010.
Groups:
- Simulation Curriculum: General surgery residents will undergo a simulation-based educational curriculum on totally extraperitoneal (TEP) hernia repair.
- Current Practice: General surgery residents will undergo training according to current practice.
Period: Overall Study
Arm/Group | Simulation Curriculum | Current Practice
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulation Curriculum | Current Practice | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (2) | 30 (3) | 30 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 17 | 18 | 35
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Participation-Corrected Operative Time
Description: Operative time was recorded with a standard stopwatch, began at the start of the operative case and ended when procedure was terminated. We realized that the operative time for poorly performing trainees could be faster than the time for more skilled trainees because the supervising surgeon would perform a greater proportion of the procedure. We calculated participation-corrected time as raw total time + the time of staff involvement: time_corrected = time_raw + (1-participation) x time_raw.
Time Frame: at first TEP procedure post-randomization; Due to surgical scheduling variability this can be anytime from 1 to 2 days following randomization to a week or two
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Simulation Curriculum | Current Practice
Number analyzed (Participants) | 26 | 24
minutes | 34.4 (8.4) | 47.5 (13.9)

2. Secondary Outcome: Operative Performance
Description: The trained observer and the staff supervising surgeon graded operative performance independently using a global rating scale, Global Operative Assessment of Laparoscopic Skills (GOALS) immediately after each case, (1 rating per case if bilateral repair). The GOALS tool has been shown to be a valid and reliable tool to measure generic laparoscopic skills in the simulated environment and in the operating room, with good agreement between live and video-review ratings. The scores range from 6 to 30, a higher score indicates greater operative performance.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simulation Curriculum | Current Practice
Number analyzed (Participants) | 26 | 24
units on a scale | 21.9 (2.7) | 18.3 (3.8)

3. Secondary Outcome: Number of Hernia Repair Subjects With Post-Operative Urinary Retention
Description: Urinary retention is the inability to empty the bladder. This is an educational study for surgeons. The participants in the study are surgeons, and the participant flow, baseline characteristics and first two outcome measures are for the surgeons. During the part of the study reported for the third outcome measure, the first surgical procedure (TEP) after randomization, each surgeon had one subject. Therefore, this outcome measure is for the hernia patients or subjects.
Time Frame: at first TEP procedure post-randomization, subjects were followed for the duration of hospital stay, an average of 1 night
Measure: Number; unit: Subjects
Arm/Group | Simulation Curriculum | Current Practice
Number analyzed (Participants) | 26 | 24
Subjects | 0 | 9

ADVERSE EVENTS:
Time Frame: Adverse events were collected on all patients during the hernia operation and postoperative until release from the hospital for first hernia repair postrandomization.
Arm/Group | Simulation Curriculum | Current Practice
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 3/26 | 24/24
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simulation Curriculum (N=26) | Current Practice (N=24)
Peritoneal tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
Epigastric vessel injury (Gastrointestinal disorders) | 1 (1) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 9 (9)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Superficial skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No